CLINICAL TRIAL: NCT00407264
Title: The Influence of Fluticasone Inhalation on Intermediate Markers of Carcinogenesis in the Bronchial Epithelium of a High Risk Population : A Double Blind Placebo-Controlled Randomised Phase II Study
Brief Title: Randomized Trial of Fluticasone in Bronchial Premalignancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: GlaxoSmithKline (Industry); The Netherlands Cancer Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FPD2001; FLU 00-02
Record Dates: First submitted 2006-11-28; First posted 2006-12-04 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Bronchogenic Carcinoma
Keywords: bronchial squamous metaplasia; bronchial squamous dysplasia
MeSH Terms: conditions — Carcinoma, Bronchogenic | interventions — Fluticasone

INTERVENTIONS:
Drug: Fluticasone propionate

SUMMARY:
The purpose of this study is to assess the efficacy of fluticasone on the development of lung cancer in smokers

DETAILED DESCRIPTION:
Bronchial epithelium exposed to cigarette smoke undergoes a series of histological changes that may ultimately lead to invasive cancer. In rats exposed to cigarette smoke inhaled corticosteroids reduce the number of lung tumors. The purpose of this study is to assess the efficacy of fluticasone on premalignant lesions in volunteers with a smoking history of >10 pack-years and patients cured of head and neck cancer or lung cancer. Participants are screened for premalignant lesions by bronchoscopy and if these are present randomised to receive a powder inhalation device containing either fluticasone 500 μg or a placebo. After 6 months, biopsies are taken from the same locations. Efficacy of treatment is assessed by reversal of metaplasia/dysplasia; secondary end-points are reversal of increased p53 immunoreactivity and hTERT expression.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* age over 18
* metaplasia index > 15%
* over 25 pack years smoking history or history of lung- or head&neck cancer
* male/female of non-childbearing potential or using approved contraception

Exclusion Criteria:

* use of inhaled/systemic corticosteroid drugs in the preceding 12 months
* contraindications for bronchoscopy/use of fluticasone
* major illness
* Baseline FEV1<1000ml
* Previous participation in clinical study
* nodules > 1cm on CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2002-02; Study Completion 2005-12

PRIMARY OUTCOMES:
Reversal of histological abnormality bronchial biopsies at 6 months

SECONDARY OUTCOMES:
Reversal of suprabasal p53 staining at 6 months
Reversal of elevated hTERT mRNA levels at 6 months
Reversal of increased KI-67 at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Egbert F Smit, MD PHD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (2):
- Netherlands (2):
  - the Netherlands Cancer Institute / Antoni van Leeuwenhoek Hospital, Amsterdam
  - VU medical center, Amsterdam

REFERENCES:
- [Background] Wattenberg LW, Wiedmann TS, Estensen RD, Zimmerman CL, Galbraith AR, Steele VE, Kelloff GJ. Chemoprevention of pulmonary carcinogenesis by brief exposures to aerosolized budesonide or beclomethasone dipropionate and by the combination of aerosolized budesonide and dietary myo-inositol. Carcinogenesis. 2000 Feb;21(2):179-82. doi: 10.1093/carcin/21.2.179. PMID 10657955
- [Background] Breuer RH, Snijders PJ, Sutedja TG, v d Linden H, Risse EK, Meijer CJ, Postmus PE, Smit EF. Suprabasal p53 immunostaining in premalignant endobronchial lesions in combination with histology is associated with bronchial cancer. Lung Cancer. 2003 May;40(2):165-72. doi: 10.1016/s0169-5002(03)00029-1. PMID 12711117